CLINICAL TRIAL: NCT00352573
Title: Values at the Bedside: A Survey of European Physicians Regarding Ethical Dilemmas in Clinical Practice
Brief Title: Ethical Dilemmas in Clinical Practice: A Survey of European Physicians
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 020247; 02-CC-0247
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Ethics
Keywords: Instrument; Physicians; Resources; Microallocation; Ethics; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Normal Volunteers: Adults over 21 years old

SUMMARY:
This study will survey a random sample of 2,100 general medicine physicians in Europe and in the U.S. about ethical difficulties they face in their practice of medicine. The participants will complete a questionnaire designed to meet the following study objectives:

* Identify the types of ethical dilemmas physicians report that they face in their practice and approaches they find helpful in responding to these situations
* Determine what ethical support physicians would find useful in dealing with ethically problematic situations
* Explore physicians experience with 'bedside rationing', due to economic or societal constraints, what procedures they forgo as a result, and what criteria they use in their rationing decisions
* Explore physicians perceptions of the equity of the health care system they work in
* Determine what interventions directed at limiting health care costs physicians would find acceptable.

Physicians in Italy, Norway, Switzerland and the United Kingdom who practice direct patient care for at least 20 percent of their time may enroll in this study.

The practice of medicine sometimes involves situations where important values come into conflict. The refusal of life-saving treatment, the concern that telling the truth could have problematic consequences, acceptable ways of facing a request to die all are examples of dilemmas that can arise in the practice of medicine. The absence of clear-cut 'right answers' to questions raised by these situations have led to the development of support services, such as ethics consultations, to help in decision-making concerning ethical problems that arise in clinical settings. Information from this survey can provide input into the continuing development of ethics support services by establishing an evidence base regarding the ethical difficulties encountered by physicians and the type of support they would consider useful in resolving these dilemmas.

DETAILED DESCRIPTION:
Ethics support services are being developed in many European countries, but the evidence base concerning the types of ethical dilemmas faced by physicians in these countries is small. The ways in which physicians respond to ethically difficult situations and the types of ethical support they would consider useful in such cases are also largely unexplored. In this study, we aim to explore the experience of physicians regarding ethical issues at the bedside in Italy, Norway, Switzerland, the UK, and the US. These are countries with very different cultural contexts, where ethics support services are in various stages of development. A better understanding of the ethical difficulties encountered by physicians in these different settings and the ways in which they respond to them would be useful locally to assist the development of support services. It would also permit intercultural comparison of the practical answers given to difficult questions for which there cannot be said that there is one right answer.

One of the ethical dilemmas faced by physicians at the bedside is the allocation of scarce resources. This is of particular interest, as it has implications that go beyond the physician-patient encounter. The choices made by physicians in situations of scarce resources not only reflect their values, but also the constraints they must work with. Knowing more about the role of those factors could be an important contribution to an evidence base for health policy.

This is an exploratory cross-sectional self-administered mailed survey of physicians in primary care in Italy, Switzerland, and the UK. The part of the survey instrument exploring physicians' experience and attitudes regarding resource allocation at the bedside will also be conducted in the U.S. The questionnaire will address the type and frequency of ethical dilemmas faced by physicians, how they approach such dilemmas, the type of ethical support they would find useful in such situations, as well as their attitudes and practices in situations of scarce resources. Data will be analyzed using descriptive statistics, factorial analysis of variance to determine factors associated with the type and frequency of ethical difficulties encountered, and logistic regression to determine factors associated with reported rationing behavior and with perception of the equity of the health care system. Independent variables used in the analysis of the last two points will also include health care systems characteristics collected from the literature. Participants will be selected on the basis of national listings. To ensure sufficient exposure to direct clinical practice, inclusion criteria will include direct patient care for at least a year and at least 20% of the participants time.

ELIGIBILITY:
* INCLUSION CRITERIA:

Physicians in Italy, Norway, Switzerland, the UK, and the U.S.

Clinical activity in Primary Care or Internal Medicine.

EXCLUSION CRITERIA:

Physicians who are not in direct patient care for at least 20% of their time.

Physicians who have not been in direct patient care for at least one year immediately prior to the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians in four European countries, Asia, Africa and the U.S.@@@
Sampling Method: Probability Sample
Enrollment: 1357 (Actual)
Dates: Start 2002-09-01 (Actual); Primary Completion 2014-07-14 (Actual); Study Completion 2014-07-14 (Actual)

PRIMARY OUTCOMES:
Explore ethical dilemmas at the bedside and micro-allocation of resources | 6 years
  Evaluate ethical dilemmas at the bedside and micro- allocation of resources via surveys after data have been collected.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Danis, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-CC-0247.html